CLINICAL TRIAL: NCT04304001
Title: Test Up Now Education Program
Acronym: TUNE-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida A&M University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: FWA00005391; U54MD007582-34A1 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-03-11 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the TUNE-UP intervention or a control group that will receive educational materials about colorectal cancer screening plus a resource list but no Community Health Advisor counseling support or cellphone / text contact like in the TUNE-UP Community Health Advisor intervention group.
Who Masked: Participant
Masking Description: Participant will complete surveys and receive mailings and not know if they are in control arm or intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Advisor (Experimental): Intervention arm participants will be scheduled to receive the Community Health Advisor intervention within 4 to 6 weeks after enrollment, a Fecal Immunochemical Test kit, a mailed targeted colorectal cancer brochure, and a follow-up telephone survey at 3- and 12-months post-intervention
  Interventions: Behavioral: Community Health Advisor
- Usual care (Active Comparator): Control group participants will receive a Fecal Immunochemical Test kit, a mailed targeted colorectal cancer brochure, and complete a follow-up telephone survey at 3- and 12-months after the mailing.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Community Health Advisor — Intervention arm participants will receive one 45-minute face-to-face meeting followed by two phone calls in one-week intervals over a period of three weeks beginning within one month following baseline survey completion. These educational activities will include the use of National Cancer Institute colorectal cancer resources and materials, including a Screen to Save media presentation, and colorectal cancer brochures. The intervention will follow a conversation guide/standard script for intervention fidelity. Community Health Advisors will take notes following each interaction to document the call length and call details. Participants will receive an additional text message reminder once a week for an additional three weeks - with instructions for participants to text "yes" to confirm they received the message - for a total of six weeks of intervention delivery. The personalized text messages will include short messages about the benefits of colorectal cancer screening.
  Arms: Community Health Advisor
Behavioral: Usual care — Control arm participants will receive a Fecal Immunochemical Test kit, a mailed targeted colorectal cancer brochure, and complete a follow-up telephone survey at 3- and 12-months after the mailing.
  Arms: Usual care

SUMMARY:
This study will test the effectiveness of an outreach strategy to increase colorectal cancer screening in African Americans. The investigators will recruit 250 African Americans ages 45-64 years who are not up-to-date with colorectal cancer screening or have never been screened, with the goal to evaluate screening knowledge, behavior, and intervention effects on colorectal cancer screening outcomes. Participants will be randomly assigned to the TUNE-UP intervention or a control group. The TUNE-UP intervention arm will utilize a community health advisor to encourage return of stool blood testing kits through cell phone outreach. The control group will receive educational materials about colorectal cancer screening plus a resource list but no community health advisor counseling support or cellphone / text contact. The primary study outcome is receipt of colorectal cancer screening (colonoscopy or Fecal Immunochemical Test) following the intervention. The secondary outcomes will include colorectal cancer screening knowledge, self-efficacy (confidence to receive colorectal cancer screening), intention to screen, and follow-up in the case of an abnormal test result. The research objective is to test the community health advisor intervention effectiveness for promoting stool blood testing as a preferred screening test in an under-screened African American population.

ELIGIBILITY:
Inclusion Criteria:

1. are 45 years to 64 years of age
2. self-identify as African American
3. have a working cellphone or telephone
4. are a resident of Florida
5. are non-adherent with colorectal cancer screening guidelines (i.e., no stool-based tests > 9 months, no colonoscopy within 9 years, and no flexible sigmoidoscopy within 4 years)
6. have no personal history of colorectal cancer, precancerous colorectal polyps, or inflammatory bowel disease (ulcerative colitis or Crohn's disease).

Exclusion Criteria:

1. under 45 years or over 64 years of age
2. do not self-identify as African American
3. do not have a working cellphone or telephone
4. not a resident of Florida
5. are adherent with colorectal cancer screening guidelines (i.e., stool-based tests < 9 months, colonoscopy within 9 years, and flexible sigmoidoscopy within 4 years) or
6. have a personal history of colorectal cancer, precancerous colorectal polyps, or inflammatory bowel disease (ulcerative colitis or Crohn's disease).

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karam Soliman, PhD, Principal Investigator — Florida A&M University
Locations (1):
- Florida A&M University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be overseen by the Principal Investigator. To facilitate sharing of data, study outcome publications from this colorectal cancer screening intervention study will provide email contact information for interested persons to obtain details on accessing de-identified data. The data sharing option will be available for at least 3 years following completion of the project, consistent with National Institutes of Health (NIH) policy on maintenance of study data.
  The investigator requesting the data will be required to submit a data request detailing the research question to be investigated, the specific variables necessary for the intended analyses, a list of individuals who will have access to the data, and proof of adequate training in the protection of human subjects for all individuals with access to data.
Supporting Information: Study Protocol, ICF
Time Frame: 3 years following completion of the project
Access Criteria: Data release will require a fully executed data sharing agreement that will place stipulations on the data that will further protect human subjects. This agreement will include the following:
  1. Requirement that the data be used for research purposes only, and not for commercial use
  2. Requirement that data will be secured using appropriate computer technology (e.g., password protected computers, firewalls)
  3. Requirement that no attempt will be made to identify any individual in the study data, and that if any identification does occur the link allowing such identification will be destroyed
  4. Requirement that data not be shared with anyone not included in the original data sharing agreement
  5. Requirement that a copy of any resulting publications be forwarded to the Principal Investigator for record-keeping purposes and for archiving as required with NIH
  6. Requirement that acknowledgment of the data source be made, as appropriate, within the investigator's publication venue

REFERENCES:
- [Derived] Luque JS, Kiros GE, Vargas MA, Ali A, Tawk R, Jackson DR, Dickey SL, Harris CM, Robinson T, Duncan B, Freeman J, Gwede CK, Wallace K. Effectiveness of a community health advisor colorectal cancer screening educational intervention on stool test completion in an African American primary care patient population: a pragmatic randomized controlled trial. BMC Glob Public Health. 2025 Jun 1;3(1):47. doi: 10.1186/s44263-025-00168-4. PMID 40450376
- [Derived] Luque JS, Matthew OO, Jackson DR, Vargas MA, Austin T, Ali A, Kiros GE, Harris CM, Tawk R, Gwede CK, Wallace K, Jean-Pierre P. Assessing the effectiveness of a community health advisor plus screen to save educational intervention on stool-based testing adherence in an African American safety net clinic population: study protocol for a randomized pragmatic trial. Trials. 2022 Feb 15;23(1):151. doi: 10.1186/s13063-022-06076-4. PMID 35168640

RESULTS

PARTICIPANT FLOW:
Groups:
- Community Health Advisor: Intervention arm participants will be scheduled to receive the Community Health Advisor intervention within 4 to 6 weeks after enrollment, a Fecal Immunochemical Test kit, a mailed targeted colorectal cancer brochure, and a follow-up telephone survey at 3- and 12-months post-intervention
  Community Health Advisor: Intervention arm participants will receive one 45-minute face-to-face meeting followed by two Community Health Advisor phone calls in one-week intervals over a period of three weeks beginning within one month following baseline survey completion. These colorectal cancer educational activities delivered by the Community Health Advisors will include the use of National Cancer Institute colorectal cancer resources and materials, including an Screen to Save media presentation, and colorectal cancer educational brochures. The intervention will follow a conversation guide/standard script for intervention fidelity. Community Health Advisors will take notes following each interaction to document the call length, deviations from the script, and tone of the call. Participants will receive an additional text message reminder once a week for an additional three weeks - with instructions for participants to text "yes" to confirm they received the message - for a total of six weeks of intervention delivery. The personalized text messages will have positive tones and include short messages about the benefits of colorectal cancer screening.
Period: Overall Study
Arm/Group | Community Health Advisor | Usual Care
Started | 58 | 57
Completed | 45 | 48
Not Completed | 13 | 9
Not completed — Lost to Follow-up | 13 | 9

BASELINE CHARACTERISTICS:
Groups:
- Community Health Advisor: Intervention arm participants will be scheduled to receive the Community Health Advisor intervention within 4 to 6 weeks after enrollment, a Fecal Immunochemical Test kit, a mailed targeted colorectal cancer brochure, and a follow-up telephone survey at 3- and 12-months post-intervention
  Community Health Advisor: Intervention arm participants will receive one 45-minute face-to-face meeting followed by two Community Health Advisor phone calls in one-week intervals over a period of three weeks beginning within one month following baseline survey completion. These colorectal cancer educational activities delivered by the Community Health Advisors will include the use of National Cancer Institute colorectal cancer resources and materials, including a Screen to Save media presentation, and colorectal cancer educational brochures. The intervention will follow a conversation guide/standard script for intervention fidelity. Community Health Advisors will take notes following each interaction to document the call length, deviations from the script, and tone of the call. Participants will receive an additional text message reminder once a week for an additional three weeks - with instructions for participants to text "yes" to confirm they received the message - for a total of six weeks of intervention delivery. The personalized text messages will have positive tones and include short messages about the benefits of colorectal cancer screening.
- Total: Total of all reporting groups
Arm/Group | Community Health Advisor | Usual Care | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.38 (5.82) | 55.07 (5.03) | 54.73 (5.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 26 | 63
  Male | 21 | 31 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 58 | 57 | 115
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 57 | 115
Colorectal Cancer Screening Knowledge Measure [Mean (Standard Deviation); unit: units on a scale] — Participants are asked four multiple choice questions and 10 True/False questions to test knowledge about colorectal cancer and colorectal cancer screening. The range of the scale is 0-14. Each answer is scored as correct or incorrect. A score of 11 to 14 is considered "high". A score of 7 to 10 is considered "average". A score less than 7 is considered "low."
  units on a scale | 9.03 (2.27) | 9.79 (2.09) | 9.41 (2.21)
Colorectal Cancer Screening Self-Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — A validated 4-item measure of colorectal cancer screening self-efficacy (alpha = 0.82) asks participants to respond using a Likert scale about colorectal cancer screening test difficulty, finding time, ease of completing the test, and scheduling the test. Total scale scores range from 1 to 4. A score of 3 to 4 is considered "low self-efficacy" and a score of 1 to 2 is considered "high self-efficacy."
  units on a scale | 1.99 (0.54) | 1.92 (0.55) | 1.95 (0.55)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Up to Date on Colorectal Cancer Screening
Description: The colorectal cancer screening measure asks about completion of colonoscopy and blood stool tests. These tests are described prior to questions about completion of each test. The first question asks when was the most recent stool blood test (> 1 year but < 2 years ago; > 2 years but not more than 5 years ago; or > 5 years). The second question asks when was the most recent colonoscopy (a year ago or less; > 1 year but < 5 years ago; > 5 years but not more than 10 years ago; or > 10 years). Colorectal cancer screening receipt will be determined based on self-report and chart review to determine screening rates for each screening modality. Those answering a "a year ago or less" for the most recent stool blood test and "less than 10 years ago" for most recent colonoscopy are considered up to date.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Advisor | Usual Care
Number analyzed (Participants) | 45 | 48
Participants | 29 | 31
Statistical Analysis 1: Comparison: Community Health Advisor vs Usual Care; For each arm, the proportion of participants who receive colorectal cancer screening by 12 months was computed. The chi-square test was used to compare the two treatment arms for screening receipt. If the proportion of participants receiving colorectal cancer screening in the intervention arm is at least 15% higher than that in the control arm, the intervention was determined to be effective; Test type: Superiority; p < 0.05, Chi-squared

2. Secondary Outcome: Colorectal Cancer Screening Knowledge Measure
Description: Participants are asked four multiple choice questions and 10 True/False questions to test knowledge about colorectal cancer and colorectal cancer screening. The range of the scale is 0-14. Each answer is scored as correct or incorrect. A score of 11 to 14 is considered "high". A score of 7 to 10 is considered "average". A score less than 7 is considered "low."
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Health Advisor | Usual Care
Number analyzed (Participants) | 45 | 48
score on a scale | 10.42 (2.01) | 9.88 (1.61)
Statistical Analysis 1: Comparison: Community Health Advisor vs Usual Care; Bivariate analyses was conducted for the knowledge scale to compare differences between the intervention and control arms. Since knowledge was a continuous variable,the values between study arms were compared using two-sample independent t-tests; Test type: Superiority; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Colorectal Cancer Screening Self-Efficacy Scale
Description: A validated 4-item measure of colorectal cancer screening self-efficacy (alpha = 0.82) asks participants to respond using a Likert scale about colorectal cancer screening test difficulty, finding time, ease of completing the test, and scheduling the test. Total scale scores range from 1 to 4. A score of 3 to 4 is considered "low self-efficacy" and a score of 1 to 2 is considered "high self-efficacy."
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Health Advisor | Usual Care
Number analyzed (Participants) | 45 | 48
score on a scale | 1.86 (0.56) | 1.98 (0.61)
Statistical Analysis 1: Comparison: Community Health Advisor vs Usual Care; Bivariate analyses was conducted for the self-efficacy scale to compare differences between the intervention and control arms. Since self-efficacy was a continuous variable, the values between study arms were compared using two-sample independent t-tests; Test type: Superiority; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed during the 2 year data collection time period.
Description: Participants only completed surveys in our study and there was no risk for adverse events from our study protocol. There were no "O" participants at risk for adverse events as this was an educational intervention study and adverse events were not monitored or assessed.All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Community Health Advisor | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The projected sample size was originally 244. Because of difficulties in recruiting this patient population of African American patients in 2 community health centers who were not up to date with colorectal cancer screening, the study was only able to recruit 115 individuals over the 2 year recruitment period. Therefore, there is smaller number of patients to analyze the effectiveness of the educational intervention, and the study is underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT04304001/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04304001/ICF_001.pdf